CLINICAL TRIAL: NCT07386288
Title: Short-term Effects of Intravenous Dexketoprofen Trometamol and Tramadol on Perfusion-Related Physiological Parameters in Renal Colic
Brief Title: Short-term Perfusion Effects: Dexketoprofen/Tramadol
Acronym: DeXTra-RC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mevlana GÜL, Asst Prof, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-16/01
Record Dates: First submitted 2026-01-20; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Renal Colic
Keywords: renal colic; emergency department; acute pain management; dexketoprofen trometamol; tramadol; tissue perfusion; end-tidal carbon dioxide
MeSH Terms: conditions — Renal Colic; Emergencies | interventions — Tramadol; dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IV Tramadol + IV Dexketoprofen (Experimental): Participants receive intravenous tramadol plus intravenous dexketoprofen trometamol for acute pain management due to renal colic. Perfusion-related physiological parameters are measured before and after administration.
  Interventions: Drug: IV Tramadol + IV Dexketoprofen Trometamol
- IV Dexketoprofen Trometamol (Experimental): Participants with renal colic receive intravenous dexketoprofen trometamol for analgesia. Perfusion-related physiological parameters are recorded at baseline and at predefined time points after administration to assess short-term effects.
  Interventions: Drug: Dexketoprofen Trometamol
- IV Tramadol (Experimental): Participants with renal colic receive intravenous tramadol for analgesia. Perfusion-related physiological parameters are recorded at baseline and at predefined time points after administration to assess short-term effects.
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Tramadol — Intravenous tramadol administered for analgesia in patients with renal colic.
  Arms: IV Tramadol
Drug: Dexketoprofen Trometamol — Intravenous dexketoprofen trometamol administered for analgesia in patients with renal colic
  Arms: IV Dexketoprofen Trometamol
Drug: IV Tramadol + IV Dexketoprofen Trometamol — Intravenous dexketoprofen trometamol and tramadol administered for analgesia in patients with renal colic
  Arms: IV Tramadol + IV Dexketoprofen

SUMMARY:
Background: Acute renal colic is a common reason for admission to the emergency department (ED) and is associated with severe pain, sympathetic activation and metabolic stress. Non-steroidal anti-inflammatory drugs (NSAIDs) and opioids are widely used for analgesia, but their short-term effects on tissue perfusion and respiratory physiology in stable patients are unclear. End-tidal carbon dioxide (EtCO₂) has been suggested as a non-invasive indicator of overall tissue perfusion, but how it behaves during analgesic treatment in stable ED patients is unclear.

Methods: This prospective, randomised study was conducted in an academic emergency department. Adult patients (aged 18-55) presenting with acute renal colic were randomised to receive an intravenous infusion of either dexketoprofen trometamol (50 mg), tramadol (100 mg), or a combination of dexketoprofen trometamol (50 mg) and tramadol (50 mg). Vital signs, oxygen saturation (SpO₂) and EtCO₂ were recorded at baseline and at 30 and 60 minutes. Arterial blood gas parameters, including lactate, were measured at baseline and after 60 minutes. The primary outcome was the change in EtCO₂ over time.

ELIGIBILITY:
Inclusion Criteria:

* A Glasgow Coma Scale score of 15
* Spontaneous respiration
* The capacity to provide informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* Chronic kidney disease,
* Known allergy to study medications,
* Chronic respiratory disease,
* Hemodynamic instability,
* Acute intoxication,
* Uncontrolled epilepsy,
* Recent monoamine oxidase inhibitor use.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change in End-Tidal Carbon Dioxide (EtCO₂) | 0, 30, and 60 minutes
  End-tidal carbon dioxide (EtCO₂) will be measured using capnography at baseline and at predefined time points following intravenous administration of tramadol and/or dexketoprofen trometamol in patients with renal colic. The primary endpoint is the change from baseline in EtCO₂.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Yakutiye Research Hospital, Yakutiye, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are not publicly available due to privacy and ethical restrictions, as they contain identifiable patient information.

REFERENCES:
- [Background] 1. Patti L, Leslie SW. Acute Renal Colic. StatPearls. Treasure Island (FL)2025. 2. Golzari SE, Soleimanpour H, Rahmani F, Zamani Mehr N, Safari S, Heshmat Y, et al. Therapeutic approaches for renal colic in the emergency department: a review article. Anesth Pain Med. 2014;4(1):e16222. https://doi.org/10.5812/aapm.16222 3. Skolarikos A, Geraghty R, Somani B, Tailly T, Jung H, Neisius A, et al. European Association of Urology Guidelines on the Diagnosis and Treatment of Urolithiasis. Eur Urol. 2025;88(1):64-75. https://doi.org/10.1016/j.eururo.2025.03.011 4. Broder JS, Oliveira JESL, Bellolio F, Freiermuth CE, Griffey RT, Hooker E, et al. Guidelines for Reasonable and Appropriate Care in the Emergency Department 2 (GRACE-2): Low-risk, recurrent abdominal pain in the emergency department. Acad Emerg Med. 2022;29(5):526-60. https://doi.org/10.1111/acem.14495 5. Morgan S. Intravenous paracetamol in patients with renal colic. Emerg Nurse. 2011;18(9):22-5. https://doi.org/10.7748/en2011.02.18.9.22.c8337 6. Holdgate A, Pollock T. Nonsteroidal anti-inflammatory drugs (NSAIDs) versus opioids for acute renal colic. Cochrane Database Syst Rev. 2004(1):CD004137. https://doi.org/10.1002/14651858.CD004137.pub2 7. Pathan SA, Mitra B, Cameron PA. A Systematic Review and Meta-analysis Comparing the Efficacy of Nonsteroidal Anti-inflammatory Drugs, Opioids, and Paracetamol in the Treatment of Acute Renal Colic. Eur Urol. 2018;73(4):583-95. https://doi.org/10.1016/j.eururo.2017.11.001 8. Cabo JJS, Miller NL. Nonopioid Pain Management Pathways for Stone Disease. J Endourol. 2024;38(2):108-20. https://doi.org/10.1089/end.2023.0266 9. Fu S, Zhang K, Gu M, Liu Z, Sun W, Xiao M. Comparative efficacy and safety of analgesics for acute renal colic: A network meta-analysis protocol. Medicine (Baltimore). 2019;98(10):e14709. https://doi.org/10.1097/MD.0000000000014709 10. Özdemir M, Çığşar Gl, Bağcıoğlu M, Çiftçi H, Günal E. Comparison of the Analgesic Effects of Intravenous Dexketoprofen, Ib

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT07386288/Prot_SAP_000.pdf